CLINICAL TRIAL: NCT02352571
Title: A Prospective, Open-label, Dose Escalation (Part A) and Cohort Expansion (Part B) Phase 1 Study to Investigate the Safety, Tolerability, and Immunogenicity and to Determine Maximum Tolerated Dose and Recommended Phase 2 Dose of GC1118 (Recombinant Human Anti-EGFR Antibody) in Patients With Advanced Solid Cancers
Brief Title: Safety Study of GC1118 (Recombinant Human Anti-EGFR Antibody) in Patients With Advanced Solid Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC1118_P1
Record Dates: First submitted 2015-01-21; First posted 2015-02-02 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-02

CONDITIONS: Neoplasm Metastasis; Gastric Cancer; Colorectal Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Stomach Neoplasms; Colorectal Neoplasms | interventions — GC1118

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single group assignment (Experimental): GC1118 recombinant human anti-EGFR antibody
  Interventions: Biological: GC1118

INTERVENTIONS:
Biological: GC1118 — For Part A, GC1118 will be administered by IV infusion once per week for 4 weeks (28-day cycles) in the dose escalation cohorts, starting 0.3mg/kg until Maximum Tolerated Dose is defined.
  For Part B, the defined MTD/RP2D of GC1118 will be administered by IV infusion once per week for 4 weeks (28-day cycles) in patients with stage IV of gastric cancer, colorectal cancer or other cancers.
  For Part C, GC1118 will be administered by IV infusion once every 2 weeks for 4 weeks (28-day cycles) in patients with all stage IV advanced solid cancers.
  Part A, Part B and Part C participants who qualify for subsequent cycles will receive continued GC1118 until evidence of progression of disease.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose(MTD)/Recommended Phase 2 Dose(RP2D) and to evaluate the safety and tolerability of GC1118 when given by intravenous (IV) infusion to patients with stage IV solid tumors.

The study will also evaluate pharmacokinetics, immunogenicity and antitumor effect of GC1118 and explore prognostic biomarkers and pharmacodynamic biomarkers.

DETAILED DESCRIPTION:
An open-label, single-arm, multi-center, phase 1, dose-escalation study will be conducted to define the MTD/RP2D, safety, PK, immunogenicity and antitumor activity of GC1118 in patients with refractory disease for whom no standard therapy is available.

This study is in three parts: a dose escalation segment (Part A), a cohort expansion (Part B) and biweekly administration(Part C). In part A, a dose escalation schema will be applied in dose level cohorts. GC1118 will be administered weekly on Study Day 1, 8, 15, and 22 of each 28-day cycle by IV infusion. Dose escalation may occur as described in the study protocol. Once the MTD has been established during Part A, the MTD cohort will be expanded in part B. And GC1118 will be administered biweekly on Study Day 1, 15 each 28-day cycle by IV infusion in part C.

Study assessments will include AE monitoring including physical examination, vital signs and clinical laboratory tests, ECG monitoring, PK analysis of serum GC1118, an assessment of potential anti-GC1118 antibody response and an exploration of potential prognostic and pharmacodynamic biomarkers.

Tumor response assessments using Study Day 36 CT/MRI scans will be performed approximately five weeks after the first GC1118 dose for each patient (Part A only). Patients with evidence of disease regression (partial or complete response or stable disease by RECIST criteria) will be allowed to continue therapy at the same dose. Subsequent cycles will consist of administration of GC1118 on Day 1, 8, 15, and 22 of each 28-day cycle with tumor evaluation every other cycle (approximately every 8 weeks) in part A,B and Day 1, 15 of each 28-day cycle with tumor evaluation every other cycle (approximately every 8 weeks) in part C.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign a written informed consent
* Nineteen (19) years of age or older
* For Part A and Part C, all stage IV advanced solid cancers For Part B, stage IV of gastric cancer, colorectal cancer or other cancer
* Cohort1: Metastatic CRC (K-RAS wild), No prior treatment with EGFR antibody therapeutics
* Cohort2: Metastatic CRC (K-RAS wild), Progressed over EGFR antibody therapeutics
* Cohort3: Advanced gastric or gastroesophageal junction cancer(EGFR++ or +++ /HER2-)
* For Part A and Part C, refractory solid tumors to conventional therapy (Progressive disease during or after previous conventional therapy)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of less than or equal to 1
* Life expectancy of greater than or equal to 3 months
* Availability of a new tumor biopsy or able to obtain unstained slides of tumor within 3 years
* For Part B, at least one measurable tumor mass by RECIST v1.1
* Acceptable laboratory parameters
* If all AEs caused by the previous anti-cancer therapies including surgery, chemotherapy and radiation therapy have recovered to CTCAE grade 1 or below (except alopecia)

Exclusion Criteria:

* Has had any major surgery or any therapy within the last 4 weeks and/or not recovered from prior therapy
* Has had chemotherapy, surgery or radiotherapy within the previous 4 weeks
* Confirmed brain metastases
* Chronic Hepatitis C or known HIV positive patients
* Liver Cirrhosis or active hepatitis B virus (HBV) carrier
* Clinically significant interstitial pulmonary disease
* Has received prior treatment with cetuximab or anti-EGFR antibody therapy is not permitted in Part B(however, allowed in Part A and Part C)
* Clinically significant cardiac disease or impaired cardiac function
* Acute or subacute intestinal obstruction or Inflammatory bowel disease
* Has had immunotherapy, chemotherapy or hormonal therapy prohibited as per study protocol
* Has participated in any study using an investigational drug during the previous 4 weeks
* Known hypersensitivity to the study drug
* History of second primary malignancy within 3 years prior to starting study treatment (excluding early gastric cancer, thyroid cancer, cervical cancer or skin cancer)
* Severe renal impairment
* Severe hepatic impairment
* Current active infection
* Known KRAS-mutation for Part A and Part C, Known KRAS-mutation for Part B or BRAF matant
* Medical or psychiatric illness that, in the opinion of the investigator, may affect compliance with scheduled visits
* Pregnant (potentially fertile patients) or lactating women
* Patients refuse to use acceptable forms of contraceptions from the time of consent through six months after the study drug administration

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Dose Limiting Toxicity (DLT) | Approx. 6 months
Frequency of Adverse Events | Approx. 6 months
Changes in safety parameters, laboratory values, vital signs and physical examinations | Approx. 6 months
  Vital sign assessment will include systolic and diastolic blood pressure, heart rate, respiration rate and temperature. Laboratory values will include hematology and clinical chemistry.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) as per Response Evaluation Criteria in Solid Tumors(RECIST) v1.1 | Approx. 6 months
Disease Control Rate (DCR) as per Response Evaluation Criteria in Solid Tumors(RECIST) v1.1 | Approx. 6 months
Progression-Free Survival (PFS) as per Response Evaluation Criteria in Solid Tumors(RECIST) v1.1 (Part B) | Approx. 6 months
Time versus plasma concentration profiles and basic PK parameters of GC1118 | Approx. 6 months
Presence of Human Anti Drug Antibody | Approx. 6 months
  Assess whether participants develop an immune response to GC1118

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Oh DY, Lee KW, Han SW, Kim JW, Shin JW, Jo SJ, Won J, Hahn S, Lee H, Kim WH, Bang YJ. A First-in-Human Phase I Study of GC1118, a Novel Anti-Epidermal Growth Factor Receptor Antibody, in Patients with Advanced Solid Tumors. Oncologist. 2019 Aug;24(8):1037-e636. doi: 10.1634/theoncologist.2019-0294. Epub 2019 Jun 4. PMID 31164456